CLINICAL TRIAL: NCT03786796
Title: Phase II Study of Olaparib in Metastatic Renal Cell Carcinoma Patients Harboring a BAP-1 or Other DNA Repair Gene Mutations (ORCHID)
Brief Title: Study of Olaparib in Metastatic Renal Cell Carcinoma Patients With DNA Repair Gene Mutations
Acronym: ORCHID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J18166; IRB00197147 (Other: JHM IRB)
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Kidney Cancer; Renal Carcinoma; Kidney Cancer Metastatic
Keywords: Olaparib
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental): Participants with metastatic renal cell carcinoma that harbor an inactivating mutation in BAP-1, ATM, BRCA1, BRCA2, PALB2, CHEK2, BRIP1, RAD51C, BARD1, CDK12, CHEK1, FANCL, PP2R2A, RAD51B, RAD51D, or RAD54L that have had prior treatment with at least one immune checkpoint inhibitor or anti-VEGF therapy with measureable disease on CT imaging according to RECIST 1.1 criteria. Participants will be initially treated with olaparib 150mg by mouth twice daily for one month. After one month of therapy, the dose will be increased to 300mg by mouth twice daily provided there are no grade 3 or greater adverse events experienced. Reassessment will occur at least monthly for toxicity. Radiological scans will be performed every 3 months to assess disease response. Treatment will be continued until clinical and/or radiographic progression according to RECIST 1.1 criteria or unmanageable toxicity requiring cessation.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib is a crystalline solid, is non-chiral and shows pH-independent solubility of approximately 0.1 mg/mL across the physiological range. Olaparib is presented for oral administration as a green, film-coated tablet containing 25 mg, 100 mg or 150 mg of drug substance. The 100 mg strength is also available as a yellow, film-coated tablet. The 25 mg, 100 mg and 150 mg strengths of olaparib tablets are composed of the same constituents. The tablet cores comprise: olaparib, copovidone, colloidal silicon dioxide, mannitol and sodium stearyl fumarate. The composition of the green tablet film coating is: hydroxypropyl methylcellulose (hypromellose), macrogol 400 (polyethylene glycol 400), titanium dioxide, iron oxide yellow and iron oxide black. The yellow tablet film coating only differs from the green film coating with the omission of iron oxide black.
  Other Names: Lynparza; AZD2281; KU-0059436; Polyadenosine 5'diphosphoribose polymerase (PARP) inhibitor

SUMMARY:
Single arm, single site, open-label Phase II study of the effects of oral olaparib in participants with metastatic renal cell carcinoma that harbor an inactivating mutation in BAP-1, ATM, BRCA1, BRCA2, PALB2, CHEK2, BRIP1, RAD51C, BARD1, CDK12, CHEK1, FANCL, PP2R2A, RAD51B, RAD51D, or RAD54L who have had prior treatment with at least one immune checkpoint inhibitor or anti-VEGF therapy. Must have measurable disease on CT imaging per RECIST 1.1 criteria.

DETAILED DESCRIPTION:
The trial will enroll up to 20 participants. Following enrollment, participants will be initially treated with olaparib 150mg by mouth twice daily for one month. After one month of therapy, the dose of olaparib will be increased to 300mg by mouth twice daily provided there are no grade 3 or greater adverse events experienced. All participants will be reassessed at least monthly for toxicity, including laboratory investigations. Radiological scans will be performed approximately every 3 months to assess for disease response. Treatment will be continued until clinical and/or radiographic progression according to RECIST 1.1 criteria or unmanageable toxicity requiring cessation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent. Provision of informed consent is required prior to any study procedures.
* Patients aged 18 years of age or older.
* Histological proof of renal cell carcinoma (both clear cell and non-clear cell allowed).
* Metastatic (AJCC Stage IV) renal cell carcinoma.
* Somatic or germline mutation in BAP-1, ATM, BRCA1, BRCA2, PALB2, CHEK2, BRIP1, RAD51C, BARD1, CDK12, CHEK1, FANCL, PP2R2A, RAD51B, RAD51D, or RAD54L as documented by a clinical CLIA-grade, tissue, saliva or blood-based genetic test.
* At least one prior treatment with an anti-angiogenic agent or immune checkpoint inhibitor.
* Any number of prior systemic therapies is allowed (cytokine, anti-angiogenic, mTOR, immune checkpoint blockage or clinical trial).
* Must have measurable disease as defined by RECIST 1.1 criteria.
* Participants must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelet count ≥ 100 x 10^9/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional ULN unless liver metastases are present in which case they must be ≤ 5 x ULN.

Note: Patients with elevations in bilirubin, AST, or ALT should be thoroughly evaluated for the etiology of this abnormality prior to entry and patients with evidence of viral infection should be excluded.

* Patients must have a creatinine clearance ≥ 40 mL/min calculated by Cockroft-Gault formula or 24 hour urine test.
* ECOG PS ≤ 1.
* Participants must have a life expectancy ≥ 16 weeks.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

Postmenopausal is defined as:

* Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments.
* Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50 years old.
* Radiation-induced oophorectomy with last menses > 1 year ago.
* Chemotherapy-induced menopause with > 1 year interval since last menses.
* Surgical sterilization (bilateral oophorectomy or hysterectomy).
* Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.

Exclusion Criteria:

* Other malignancy unless curatively treated with no evidence of disease for ≥ 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma. Patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy > 3 years prior to registration, and that the patient remains free of recurrent or metastatic disease.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Breast feeding women.
* Use of any prohibited concomitant medications within the prior 2 weeks.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Participation in another clinical study with an investigational product during the last 2 weeks.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment.
* Any previous treatment with PARP inhibitor, including olaparib.
* Resting ECG with QTc > 500 ms and/or indication of uncontrolled cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, electrolyte disturbances, etc.), or patients with congenital and/or family history of long QT syndrome.
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks. During the study, if co-administration of a strong or moderate inhibitor is required because there is no suitable alternative medication, exception to this criterion may be allowed with a suitable dose reduction of olaparib.
* Concomitant use of known strong CYP3A inducers (e.g. phenobarbital, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital or enzalutamide and 3 weeks for other agents.
* Persistent toxicities (> Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Known hypersensitivity to olaparib or any of the excipients of the product.
* Known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* No packed red blood cells and/or platelet transfusions within the last 28 days prior to study entry.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response or Stable Disease to Olaparib Therapy at Six Months | 6 months post-intervention
  Complete response (CR) or partial response (PR) at any time on study or stable disease (SD) after 6 months of Olaparib treatment, based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Safety of Olaparib Therapy As Determined by the Number of Adverse Events | 2 years
  Number of Adverse Events, Grade 3 or higher as defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Median Progression-Free Survival to Olaparib Therapy | 2 years
  Number of months from the time of initiation on Olaparib therapy until radiographic progression or death, whichever comes first while enrolled on the study, based on RECIST 1.1 criteria.
Rate of Objective Response to Olaparib Therapy | 2 years
  Number of participants with best overall response (complete response (CR) or partial response (PR)) at anytime on study.

OTHER OUTCOMES:
Reversion Mutations in Circulating Tumor DNA (ctDNA) at Clinical Progression | 2 years
  Number of incidences of reversion mutations in circulating tumor DNA (ctDNA) at time of clinical progression.

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Markowski, MD, Ph.D, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No